CLINICAL TRIAL: NCT05792215
Title: Dental Practitioners' Knowledge, Attitude, and Practice (KAP) in Cairo and Riyadh Regarding Caries Risk Assessment and Management: A Cross-Sectional Study
Brief Title: KAP of Dental Practitioners Regarding CRA
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed Saqer Saeed Almutairi, Principal Investigator, Cairo University
Other Study IDs: KAP Regarding CRA
Record Dates: First submitted 2023-03-18; First posted 2023-03-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Caries,Dental; Tooth Decay; Tooth Diseases
Keywords: Caries Risk Assessment; Caries Prevention; General Practitioners
MeSH Terms: conditions — Dental Caries; Tooth Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the knowledge, attitude, and practice of a group of dental practitioners from Cairo and Riyadh regarding caries risk assessment and management.

DETAILED DESCRIPTION:
Dental caries is a preventable major public health disease affecting people of all ages and substantially impacting overall health. Caries remain the single most common chronic childhood disease. Dental caries is a dynamic and complex process. Several variables influence the occurrence of dental caries, including oral flora, saliva flow and composition, and lifestyle. Dental caries development can be primary (new carious lesion) or secondary (lesion progression or reactivated carious lesions).

There has been much progress over the past several decades in the prevention of dental caries, shifting from the management of dental caries from a "surgical approach" to a "medical prevention strategy", based on a better understanding of the caries disease process.

Caries Risk Assessment (CRA) is a significant part of successfully applying the minimum intervention dentistry philosophy in managing dental caries. As recommended by AAPD, Dental caries-risk assessment should be a routine component of new and periodic examinations by oral health and medical providers. Therefore, this study aims to assess the knowledge, attitude, and practice of a group of dental practitioners from Cairo and Riyadh regarding caries risk assessment and management.

Benefits to Practitioner:

* Increasing awareness of the importance of CRA practices.
* Implementing a positive attitude regarding CRA and management.
* Improve practices toward CRA

Benefits to Patient:

* Increasing the awareness and knowledge of early caries prevention by dentists.
* Increasing awareness about Caries Risk Assessment and management.

Benefits to Community:

• Increasing the knowledge and awareness of the community regarding preventive dentistry and the importance of primary prevention

ELIGIBILITY:
Inclusion Criteria:

* Licensed Egyptian and Saudi general dentists.

Exclusion Criteria:

* Undergraduate dental students
* Dental specialists
* Dentists who refused to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All licensed Egyptian and Saudi general dentists
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge, Attitude, and Practice of Dental Practitioners in Cairo and Riyadah | 1 year
  Questionnaire
  The questionnaire is composed of the following sections:
  (A) Sociodemographic data including participants' age, gender, qualification, experience years, place of practice, and the number of pediatric patients they see every week.
  (B) Participants' knowledge of caries risk assessment indicators.
  Section (B) will contain binary questions (true and false)
  (C) Participants' attitudes and knowledge related to caries risk assessment and management.
  section (C) will contain three-point Likert scale (''Agree'', ''Disagree'' and "Neither agree nor disagree")
  (D) Barriers in caries risk assessment and management practices.
  Section (D) will contain a four-point Likert-type scale (always, often, sometimes, and never.)

CONTACTS AND LOCATIONS:
Overall Officials: Gihan M Abuelniel, Professor, Study Chair — Professor